CLINICAL TRIAL: NCT01038752
Title: Combination of Non-Cytotoxic Suramin With Docetaxel and Carboplatin in Chemo-Naive Non-small Cell Lung Cancer (NSCLC): A Randomized Single-Blind Placebo-Controlled Phase II Study
Brief Title: Evaluation of Non-cytotoxic Suramin as a Chemosensitizer in Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Optimum Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Optimum-Suramin-1
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; suramin; lung cancer; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Suramin; Docetaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suramin (Experimental): This group will receive the combination of non-cytotoxic suramin with docetaxel and carboplatin.
  Interventions: Drug: Suramin Drug:Docetaxel Drug: Carboplatin
- Standard of care (Placebo Comparator): This group will receive placebo with docetaxel and carboplatin.
  Interventions: Drug: Placebo Drug: Docetaxel Drug: Carboplatin

INTERVENTIONS:
Drug: Suramin Drug:Docetaxel Drug: Carboplatin — Suramin dosage will be determined by nomogram and administered over 30 minutes. Suramin is followed by docetaxel (56 mg/m2, administered over 1 hour), followed by carboplatin (dosage calculated by Calvert equation to have a target AUC of 6, administered over 1 hour).
  Other Names: CI-1003; PD 002927-0015F; NSC 34936; Bayer 205; Germanin; Metaret; Taxotere; Paraplatin
  Arms: Suramin
Drug: Placebo Drug: Docetaxel Drug: Carboplatin — Placebo (100 ml of 0.9% sodium chloride or 5% dextrose in water) will be administered over 30 minutes, followed by docetaxel (75 mg/m2, administered over 1 hour), followed by carboplatin (dose calculated by Calvert equation to have a target AUC of 6, administered over 1 hour).
  Other Names: Taxotere; Paraplatin
  Arms: Standard of care

SUMMARY:
The purpose of this study is to evaluate the benefit of adding suramin at a non-cytotoxic dose to carboplatin and docetaxel regimen in the treatment of chemo-naïve patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
The primary objective is to determine the progression free survival for patients with stage III B with malignant pleural effusion or Stage IV NSCLC treated with docetaxel and carboplatin with or without suramin.

The secondary objectives are to compare median overall survival rate, compare overall response rate of patients in both arms, assess toxicity of suramin with docetaxel and carboplatin, determine whether pre-treatment bFGF levels correlate with survival, to determine whether survival benefit from suramin is associated with M phase entry in peripheral blood lymphocytes, and to determine whether adding suramin to docetaxel and carboplatin produces greater survival benefits in African-American patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven on-small cell lung cancer (NSCLC), including squamous cell carcinoma.
* Newly-diagnosed stage IIIB with malignant pleural effusion, stage IV or recurrent disease.
* Known central nervous system metastases if patients are asymptomatic and have completed whole brain or stereotactic radiation at least 2 weeks prior or surgery at least 4 weeks prior to starting treatment on this protocol. Must be off dexamethasone at the time of starting treatment.
* Must have completed radiotherapy at least two weeks prior to registration. Prior radiation therapy is eligible if patient has a measurable lesion that has not been irradiated.
* Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (RECIST criteria).
* Lesions that are not considered measurable include the following:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
  * Tumor lesions situated in a previously irradiated area
* ECOG performance status of 0-1.
* Life expectancy ≥ 3 months.
* Adequate bone marrow function, absolute neutrophil count ≥1,500/mm3, hemoglobin ≥9.9 gm/dl, and platelet count ≥100,000/mm3.
* Adequate liver function defined as bilirubin ≤ 1x upper level of the institutional normal (ULIN). AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the two values (AST or ALT) should be used. See protocol.
* Must have adequate renal function defined as serum creatinine ≤ 2.0 mg/dl or calculated creatinine clearance ≥ 60 ml/min for patients with creatinine levels above 2.0 mg/dl.
* Must have recovered from uncontrolled intercurrent illness, including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Use of adequate contraception (hormonal or barrier method of birth control) for the duration of study participation and continued for at least three months after completing treatment. Non-pregnant status will be determined in all women of childbearing potential.
* Age > 18.
* Patients must have given written informed consent.
* Entry to this study is open to both men and women and to all racial and ethnic subgroups. The goal is to accrue a minimum of 44 patients of African-American ancestry and a maximum of 120 non-African-American patients. Classification of patient race and ancestry will be based on patient's self-identification on the consent form for the clinical trial.

Exclusion Criteria:

* History of severe hypersensitivity reaction to Docetaxel or other drugs formulated with polysorbate 80.
* Grade 3 or 4 neuropathy.
* Women who are pregnant or breast-feeding.
* Prior chemotherapy or biologic therapy (e.g., erlotinib) for NSCLC including neoadjuvant or adjuvant chemotherapy.
* Currently active second malignancy other than non-melanoma skin cancer. Currently active malignancy does not include prior malignancy treated with therapy and considered to have less than 30% risk of relapse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 164 subjects were expected to be enrolled in this study; however, only a total of 14 subjects were enrolled at two active sites. Site 001 (Virginia Commonwealth University) enrolled 4 subjects and site 002 (Cook County) enrolled 10 subjects for a total of 14 subjects.
Groups:
- Suramin: This group will receive the combination of non-cytotoxic suramin with docetaxel and carboplatin.
  Suramin, Docetaxel, Carboplatin: Suramin dosage will be determined by nomogram and administered over 30 minutes. Suramin is followed by docetaxel (56 mg/m2, administered over 1 hour), followed by carboplatin (dosage calculated by Calvert equation to have a target AUC of 6, administered over 1 hour).
- Standard of Care: This group will receive placebo with docetaxel and carboplatin.
  Placebo, Docetaxel, Carboplatin: Placebo (100 ml of 0.9% sodium chloride or 5% dextrose in water) will be administered over 30 minutes, followed by docetaxel (75 mg/m2, administered over 1 hour), followed by carboplatin (dose calculated by Calvert equation to have a target AUC of 6, administered over 1 hour).
Period: Overall Study
Arm/Group | Suramin | Standard of Care
Started | 8 | 6
Completed | 3 | 1
Not Completed | 5 | 5
Not completed — Tumor Progression | 2 | 2
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Suramin: This group will receive the combination of non-cytotoxic suramin with docetaxel and carboplatin.
  Suramin + Docetaxel + Carboplatin: Suramin dosage will be determined by nomogram and administered over 30 minutes. Suramin is followed by docetaxel (56 mg/m2, administered over 1 hour), followed by carboplatin (dosage calculated by Calvert equation to have a target AUC of 6, administered over 1 hour).
- Standard of Care: This group will receive placebo with docetaxel and carboplatin.
  Placebo + Docetaxel + Carboplatin: Placebo (100 ml of 0.9% sodium chloride or 5% dextrose in water) will be administered over 30 minutes, followed by docetaxel (75 mg/m2, administered over 1 hour), followed by carboplatin (dose calculated by Calvert equation to have a target AUC of 6, administered over 1 hour).
- Total: Total of all reporting groups
Arm/Group | Suramin | Standard of Care | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Non-small cell lung cancer (NSCLC) Disease Stage at Entry [Number; unit: participants] — Stage I: The cancer is confined only to the lungs.
  Stage II: The cancer is in the lung and nearby lymph nodes.
  Stage III: Cancer is found in the lung and in the lymph nodes in the middle of the chest. There are two subtypes:
  * A: Cancer has spread only to lymph nodes on the same side of the chest where the cancer started.
  * B: Cancer has spread to the lymph nodes on the opposite side of the chest, or above the collar bone.
  Stage IV: When the cancer has metastasized to both lungs, to fluid in the area around the lungs, or to another part of the body, such as the liver or other organs.
  participants
    IIIB | 1 | 0 | 1
    IV | 7 | 6 | 13
Non-small cell lung cancer (NSCLC) Disease Type [Number; unit: participants]
  Squamous | 2 | 2 | 4
  Nonsquamous | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival for Participants With Stage IIIB/IV NSCLC Per RECIST Criteria
Description: Insufficient data
Time Frame: Patients will be followed every 2 months for the first 6 months following the last cycle of treatment, every three months for the next year, and every 6 months thereafter.
Population: Because 6 of 14 participants were lost to follow up before progression, analysis was not performed.
Arm/Group | Suramin | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival of Participants
Description: Insufficient Data
Time Frame: First treatment date to date of death
Population: Because 6 of 14 participants were lost to follow up before progression, analysis was not performed.
Arm/Group | Suramin | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Response Rate (Complete Response + Partial Response) of Participants
Description: Insufficient data
Time Frame: Tumor assessment at every other cycle
Population: Because 6 of 14 participants were lost to follow up before progression, analysis was not performed.
Arm/Group | Suramin | Standard of Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Toxicity of Combination of Non-cytotoxic Suramin With Docetaxel and Carboplatin.
Description: Insufficient data.
Time Frame: Day 1 of each cycle; end of treatment visit; at follow-up.
Population: Because 6 of 14 participants were lost to follow up before progression, analysis was not performed.
Arm/Group | Suramin | Standard of Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pre-treatment bFGF Levels Correlation With Survival.
Description: Insufficient data.
Time Frame: Before first treatment
Population: Because 6 of 14 participants were lost to follow up before progression, analysis was not performed.
Arm/Group | Suramin | Standard of Care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Survival Benefit From Non-cytotoxic Suramin Association With Reduced M-phase Entry in Peripheral Blood Lymphocytes
Description: Insufficient data.
Time Frame: Randomization date
Population: Because 6 of 14 participants were lost to follow up before progression, analysis was not performed.
Arm/Group | Suramin | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: To Determine Whether Adding Non-cytotoxic Suramin to Docetaxel and Carboplatin Produces Survival Benefits in African-American Patients.
Description: Insufficient data.
Time Frame: Randomization date to date of death
Population: Because 6 of 14 participants were lost to follow up before progression, analysis was not performed.
Arm/Group | Suramin | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: To Determine Whether Adding Non-cytotoxic Suramin to Docetaxel and Carboplatin Produces Greater Survival Benefits in African-American Patients Compared to Non-African-American Patients.
Description: Insufficient data.
Time Frame: Randomization date to date of death
Population: Because 6 of 14 participants were lost to follow up before progression, analysis was not performed.
Arm/Group | Suramin | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Suramin | Standard of Care
Serious Adverse Events (participants affected / at risk) | 3/8 | 0/6
Other Adverse Events (participants affected / at risk) | 6/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suramin (N=8) | Standard of Care (N=6)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated to the treatment and determined to be caused by disease progression.
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Unrelated to the treatment and determined to be caused by disease progression.
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) — Unrelated to treatment or cancer and possibly result of an infection.
Altered mental status (Psychiatric disorders) | 1 (1) | 0 (0) — Attributed to acute ischemia and not related to treatment.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Attributed to the progression of disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suramin (N=8) | Standard of Care (N=6)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 6 (23)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Fatigue/asthenia (General disorders) | 5 (11) | 5 (22)
Thrombosis (Vascular disorders) | 3 (6) | 0 (0)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (5) | 1 (4)
Nausea (General disorders) | 5 (9) | 1 (1)
Vomiting (General disorders) | 3 (4) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (8)
Mayalgias/Arthralgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Constipation (General disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0)
Abdominal Pain/Cramps (General disorders) | 2 (2) | 0 (0)
Hypersensitivity/Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0)
Transaminitis (Hepatobiliary disorders) | 0 (0) | 0 (0)
Hearing Loss/Tinnitus (General disorders) | 0 (0) | 1 (1)
Fluid Retention/Edema (General disorders) | 1 (1) | 2 (4)
Peripheral Neuropathy (Nervous system disorders) | 1 (1) | 1 (2)
Seizures (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to the loss of follow-up of 6 of 14 participants before progression and slow accrual. Due to the resulting small numbers, no analysis was attempted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No